CLINICAL TRIAL: NCT05466331
Title: Drug Injection Surveillance and Care Enhancement for Rural Northern New England (UH3)
Brief Title: Rural New England Health Study (Phase 2)
Acronym: DISCERNNE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baystate Medical Center (Other)
Collaborators: Tufts University (Other); University of New Hampshire (Other); University of Vermont (Other); Dartmouth-Hitchcock Medical Center (Other); Better Life Partners Inc (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH19-166; UH3DA044830 (NIH)
Record Dates: First submitted 2022-06-13; First posted 2022-07-20 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Hepatitis C; Opioid Use Disorder; IV Drug Usage
MeSH Terms: conditions — Hepatitis C; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Tele-HCV Care (Experimental): Direct Acting Antiviral (DAA) treatment for HCV on a mobile van via telemedicine
  Interventions: Other: Mobile Tele-HCV Care
- Enhanced Usual Care (Active Comparator): Referral with care navigation to a local or regional HCV treatment provider
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Other: Mobile Tele-HCV Care — Study participants receive HCV care via telemedicine. Telemedicine appointments are performed on a mobile van.
  Arms: Mobile Tele-HCV Care
Other: Enhanced Usual Care — Study participants are referred to a clinician in their area for HCV care.
  Arms: Enhanced Usual Care

SUMMARY:
This study will integrate mobile hepatitis C virus (HCV) testing and treatment with expanded syringe access in order to improve uptake of HCV testing and treatment, and reduce syringe sharing behavior in rural northern New England. The intervention aims to reach rural opioid injectors with HCV and to fill service gaps identified around access to syringe services and HCV testing and treatment, while limiting the burden on local partners. If effective, this mobile model of HCV telehealth integrated with syringe services will provide a promising approach for local public health authorities seeking to curb opioid injection, syringe sharing and HCV rates in rural America, and reduce the risk environment for HIV outbreaks in those communities.

DETAILED DESCRIPTION:
This study will employ a randomized, parallel-group design to determine the best strategy for mobile testing-and-treatment of rural opioid users for HCV. This Type 1 hybrid effectiveness-implementation study will examine the effectiveness of a model of mobile telemedicine service delivery integrated into rural harm reduction programming. The model aims to reach rural opioid injectors who are living with HCV and to fill service gaps identified in previous work around access to syringe services and HCV testing and treatment. Working closely with local harm reduction agencies, this study will employ a mobile van to expand antibody and viral load testing for HCV, distribute syringes in rural communities with poor access to brick-and-mortar syringe service providers, and provide HCV telemedicine treatment. The study will also replicate prior validation of the accuracy of dried blood spot (DBS) testing for HCV viral load as a potential strategy to address limited access to effective phlebotomy. All consenting volunteers with HCV antibody present will receive HCV viral load and liver elastography results, and, if current HCV carriers, initial vaccination for HBV and/or HAV. Participants with current HCV will be randomized to one of two intervention arms for HCV work-up and care.

ELIGIBILITY:
Inclusion Criteria:

1. Current or past history of drug injection;
2. Health insurance that will cover HCV medications (study staff will work with those who are eligible but have not signed up for insurance prior to study enrollment)
3. Lives in one of the study counties in NH and VT, and plans to remain in the study region for the next 12 months;
4. Age 18 years or older;
5. Speaks English;
6. Capacity to voluntarily provide informed consent;
7. Will accept randomized assignment, and participate in follow-up over 12 months;
8. Will provide releases to access community medical records;
9. Will provide names and contact information of at least 3 persons for re-contact purposes;
10. Not previously treated for HCV;
11. Not pregnant or trying to conceive;
12. HCV antibody positive on point-of-care rapid test.

Exclusion Criteria:

1. Unable to obtain venous blood sample for mandatory laboratory testing
2. HCV viral load undetectable
3. Hepatitis B surface antigen (HBsAg) positive;
4. Significant renal failure (eGFR 30 mL/min/1.73m2 or less, or end-stage renal disease requiring dialysis);
5. Decompensated cirrhosis, as manifested by liver fibrosis on elastography (FibroScan) and/or Fibrosure blood test plus at least one of the following symptoms:

i. Observed jaundice (yellowing of the eyes and skin) ii. Self-reported increasing abdominal size (ascites) and leg edema iii. Observed periods of confusion consistent with encephalopathy iv. Self-reported history of gastrointestinal bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Treatment initiation | 16 weeks post-enrollment
  Proportion of participants who initiate DAA treatment
Sustained virologic response | 12 weeks post-treatment
  Proportion of participants who achieve sustained virologic response at 12 weeks post-treatment. Sustained virologic response means that RNA from hepatitis C virus is not detectable in blood samples.
Syringe sharing | 24 weeks post-treatment
  Proportion of participants who report no syringe sharing in the prior 30 days at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Friedmann, MD, MPH, Principal Investigator — Baystate Medical Center; Thomas J Stopka, PhD, MHS, Principal Investigator — Tufts University
Locations (3):
- United States (3):
  - Mobile Study Van, Keene, New Hampshire
  - Mobile Study Van, Bennington, Vermont
  - Mobile Study Van, Brattleboro, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Friedmann PD, Wilson D, de Gijsel D, Nolte K, Dejace J, Hoskinson R Jr, Del Toro-Mejias L, Bianchet E, Dowd P, Soares WE 3rd, Stopka TJ. Mobile Telemedicine for Treating Chronic Hepatitis C Among Rural People Who Inject Drugs: A Randomized Clinical Trial. JAMA Netw Open. 2026 Jan 2;9(1):e2555125. doi: 10.1001/jamanetworkopen.2025.55125. PMID 41587029